CLINICAL TRIAL: NCT05663385
Title: Alveolar Ridge Preservation With a Xenograft (Bio-Oss® Collagen) and a Collagen Matrix (Mucograft® Seal) or a Free Connective Tissue Graft Versus Spontaneous Healing:A 5-year Follow up
Brief Title: Mucograft Seal in ARP Follow-up
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Dr. Justin Pijpe, Assistent Professor, Erasmus Medical Center
Other Study IDs: NL82943.078.22
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Dental Implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Rationale: Early implant placement with alveolar ridge preservation (ARP) using either a collagen matrix or a palatal graft rendered similar esthetic, clinical and PROMs to early implant placement without ARP, up to 1 year after functional loading.

Objective: The aim of this study is to evaluate esthetic and clinical outcomes and patient satisfaction following single-tooth replacement in the anterior maxilla in patients treated with a xenograft and a collagen matrix or a free connective tissue graft versus spontaneous healing 5 years after loading

Study design: prospective observational study with 5-year follow-up

Intervention (if applicable): not applicable

Main study parameters/endpoints: Comparison of the level of the buccal marginal gingiva (midfacial mucosa level) between ARP versus spontaneous healing

Secondary parameters/endpoint: Peri-implant esthetic score (PES) and white esthetic score (WES), complications, implant survival; and success, Plaque Index, Modified bleeding index, Gingival Index, Probing Depth, PROMs, bone and soft tissue volumetric dimensional changes.

DETAILED DESCRIPTION:
Replacement of a single tooth in the esthetic zone is a demanding procedure. For optimal esthetic results, no deficiency in both bone and soft tissue is acceptable. Immediately after tooth extraction, the alveolar ridge undergoes horizontal and vertical bone loss. This negatively influences the soft tissue contours, and thus esthetic outcome. Although immediate placement of an implant after extraction leads to acceptable esthetic results, there is an increased risk of mucosal recession due to the lack of adequate soft tissue. Early implant placement, 4 to 8 weeks after extraction, may offer advantages in terms of soft and hard tissue preservation. The main goals when treating the extraction socket in the esthetic zone is to preserve as much as possible existing soft and hard tissue volume as possible for future implant placement. Landsberg described a modified ridge preservation technique called "socket seal surgery" where flap elevation is avoided and it combines both bone and soft tissue grafting prior to implant placement. Closing the extraction site from the oral cavity using a thick epithelized palatal graft enables optimal ridge preservation immediately after tooth extraction. Jung showed that the application of a slowly resorbing biomaterial (BioOss Collagen®, Geistlich) into an extraction socket, covered with an autogenous palatal soft tissue punch graft resulted in a high predictability and reliability for a good esthetic result for future (early) implant placement. Although a soft tissue graft is a relatively easy procedure, patient morbidity is often associated with the second surgical site. An artificial socket seal might prevent donor morbidity associated with soft tissue grafts. A critical determinant for stable esthetic long-term outcomes is integrity and stability of the facial bone wall. The application of a biomaterial into an extraction socket, covered with a collagen matrix or a soft tissue graft, resulted in less vertical and horizontal changes of the alveolar ridge 6 months after extraction. Although there seems to be no difference in the long term change of the buccal soft tissue contour and alveolar ridge between a collagen matrix and an autogenous soft tissue punch graft, there is a lack in data concerning the difference in esthetic outcome between these two methods in early implant placement. Therefore, we evaluated esthetic and clinical outcomes and patient satisfaction following single-tooth replacement in the anterior maxilla in patients treated with alveolar ridge preservation(ARP) with a xenograft (Bio-Oss® Collagen) and a collagen matrix (Mucograft® Seal) or a free connective tissue graft versus spontaneous healing up to 1 year after functional loading (MEC-2015-016;NL49965.078.14). This study showed that ARP using a xenogeneic bone substitute covered with a collagen matrix or a palatal graft, resulted in less bone resorption and fewer bone augmentation procedures at early implant placement compared to spontaneous healing. One year after functional loading, there was no difference in clinical and esthetical outcomes and similar PROMS between the three treatment modalities. In order to achieve optimal esthetic results, both the bone and soft tissue have to be preserved as good as possible. Not much is known about the long term stability of ARP compared to spontaneous healing and PROMs.

ELIGIBILITY:
Inclusion Criteria:

* All patients previously included in the above mentioned RCT.

Exclusion Criteria:

* Patients treated with radiotherapy during follow-up in the head-and-neck region or current chemotherapy; disability (mental and/or physical) to maintain basic oral hygiene procedures.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients were included in a prospective randomized clinical trial comparing alveolar ridge preservation with a xenograft and a collagen matrix or a free connective tissue graft versus spontaneous healing (MEC-2015-016;NL49965.078.14).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
buccal marginal gingival level | 5 year
  1. Is the buccal marginal gingival level (midfacial mucosa level) of implants treated post-extraction with a bone substitute material (BioOss® Collagen) and a collagen matrix (Geistlich Mucograft® Seal) (Group A) or covered with a palatal graft (Group B) more favorable then the buccal marginal gingiva in spontaneous healing (Group C) up to 5 year after functional loading?

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Mc, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No